CLINICAL TRIAL: NCT00051519
Title: Screening HIV-Infected Subjects for Vaccine Research Studies
Brief Title: Screening HIV-Infected Patients for Vaccine Studies
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030079; 03-I-0079
Record Dates: First submitted 2003-01-10; First posted 2003-01-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-25

CONDITIONS: HIV Infection
Keywords: HIV; AIDS; Vaccine; HIV-positive; Therapy
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; HIV Seropositivity

SUMMARY:
This screening study will evaluate potential study volunteers with HIV infection to see if they are suitable candidates for trials of experimental vaccines against HIV (therapeutic), and against other infections (preventive).

* Preventive vaccines against other infections. Preventive vaccines prevent a person from getting a disease. Preventive vaccines have been developed for many diseases, including, for example, whooping cough, measles, mumps, influenza, and hepatitis B. Some preventive vaccines may also prevent a disease from taking hold if given immediately after infection, such as vaccines for rabies, smallpox and hepatitis.
* Therapeutic vaccines against HIV. Therapeutic vaccines are intended to treat someone who has already been infected, with the goal of controlling the disease or preventing it from causing severe illness. As yet, there are no therapeutic vaccines for any diseases.
* Vaccines against other infections. Vaccines to prevent other infections besides HIV may need to be tested separately in people with HIV infection because the immune system works differently when HIV infection is present.

HIV-infected patients 18 years of age or older may be eligible for this screening study. Women who are pregnant or breast feeding may not participate.

Participants will be screened with the following:

* A health history, including questions about sexual activity and drug use;
* Physical examination, including blood and urine tests;
* HIV testing to confirm HIV infection;
* Pregnancy test for premenopausal women;
* PPD test for tuberculosis for those who have not been tested in the previous 6 months.

Candidates who meet the requirements for investigational vaccine studies will be invited to participate in a study. Those who do not begin a study within 1 month of the screening tests may need to repeat some tests for continued consideration. In addition, some studies require repeated measures of CD4 counts and viral load over a period of a few months.

DETAILED DESCRIPTION:
Study Design: The purpose of this protocol is to screen potential study volunteers with HIV infection to determine if they are suitable candidates for vaccine trials. Screening will be primarily for HIV vaccine trials, but may also be for screening HIV-infected adults to participate in trials of other kinds of vaccine studies that will be enrolling HIV-infected subjects. All work will be conducted at the National Institutes of Health. HIV-infected volunteers will be recruited and screened. This protocol will be used to determine if the volunteers meet eligibility requirements for participation in trials of vaccines in HIV-infected subjects.

Subjects: Approximately 1,000 adults with HIV infection.

Study Plan: Subjects are evaluated for eligibility to participate in a vaccine trial and receive counseling on HIV-related issues. Women receive counseling on avoidance of pregnancy during a clinical trial. If it is determined that the volunteer might be eligible for a vaccine trial, additional information about trial options will be provided by telephone, mail and/or visits with a study coordinator.

Study Duration: Approximately six months for each subject.

Study Evaluations: Evaluations usually include history and physical examinations and CBC, differential, platelets, PT/PTT, chemistry panel, urinalysis, pregnancy test for women of reproductive potential, hepatitis B surface antigen, hepatitis C antibody, RPR, ELISA and Western blot for HIV, anti-dsDNA, quantitative immunoglobulins, adenovirus serology and T cell subsets (CD4/CD8). However, only those evaluations needed to determine eligibility for a particular vaccine study will be completed. Blood will also be collected for storage. If needed for eligibility in a particular vaccine study, a PPD will be administered unless subject has documentation of a negative PPD within six months prior to enrollment. In addition, other standard clinical evaluations may be done if needed to determine eligibility for a particular vaccine study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 years or older

HIV-infected, confirmed by ELISA and Western blot

Willing to participate for the planned duration of the study (6 months or longer)

Able and willing to give informed consent

Agree to have blood stored for future studies related to HIV, the immune system, vaccine response and/or other medical conditions

EXCLUSION CRITERIA:

Women who are known to be pregnant or breast feeding

Clinically significant medical history, physical examination or laboratory test results that preclude participation in a clinical trial.

A condition requiring medication that affects the immune response to a vaccine such as oral and parenteral corticosteroids, hydroxyurea, interleukin-2 or other immune modulators.

A condition in which repeated blood draws or injections poses more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access.

A condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being

A condition in which signs or symptoms could be confused with reactions to vaccine

Active participation in other experimental treatment studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2003-01-09; Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States